CLINICAL TRIAL: NCT02140450
Title: Short Term Intraocular Pressure Fluctuations After Intravitreal Bevacizumab Injection: the Effect of Pretreatment With Antiglaucoma Agents
Brief Title: Effect of Antiglaucoma Agents on Short Term Intraocular Pressure Fluctuations After Intravitreal Bevacizumab Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasser Shoeibi, Assistant Professor of Ophthalmology, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 910292
Record Dates: First submitted 2014-05-09; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Intraocular Pressure Change in Intravitreal Injection
Keywords: intraocular pressure, intravitreal injection, short term
MeSH Terms: interventions — Timolol; Brimonidine Tartrate; Acetazolamide; Mannitol; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Timolol (Active Comparator): Timolol eyedrop, 2 drops 5 minutes apart, 1-2 hours before intravitreal injection
  Interventions: Drug: Timolol
- Brimonidine (Active Comparator): Brimonidine eyedrop, 2 drops 5 minutes apart, 1-2 hours before intravitreal injection
  Interventions: Drug: Brimonidine
- Acetazolamide (Active Comparator): Acetazolamide tablet, 2 tabs, 2 hours before intravitreal injection
  Interventions: Drug: Acetazolamide
- Mannitol (Active Comparator): Intravenous mannitol, 1.5 gram/kg, 1 hour before intravitreal injection
  Interventions: Drug: Mannitol
- Placebo (Sham Comparator): Artificial tears, 2 drops, 1-2 hours before intravitreal injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Timolol — 2 drops of timolol, 10 minutes apart, 1-2 hours before intravitreal injection
  Other Names: Timoptic
  Arms: Timolol
Drug: Brimonidine — Brimonidine eyedrop, 2 drops 5 minutes apart, 1-2 hours before intravitreal injection
  Other Names: Alphagan
  Arms: Brimonidine
Drug: Acetazolamide — Acetazolamide tablet, 2 tabs, 2 hours before intravitreal injection
  Other Names: Diamox
  Arms: Acetazolamide
Drug: Mannitol — Intravenous mannitol, 1.5 gram/kg, 1 hour before intravitreal injection
  Arms: Mannitol
Drug: Placebo — Artificial tears, 2 drops, 1-2 hours before intravitreal injection
  Other Names: Sham
  Arms: Placebo

SUMMARY:
To assess the effect of prophylactic antiglaucoma agents in prevention of acute intraocular pressure rise after intravitreal injection.

DETAILED DESCRIPTION:
Acute intraocular pressure elevation after intravitreal injection of bevacizumab was proven.Acute intraocular pressure elevation most probably is volume related and long term intraocular pressure elevation relates to pharmacologic features of the medications which results in anatomic changes in the angle of anterior chamber.Numerous studies found an intraocular pressure elevation right after the injection and quick normalization within maximally 30 minutes.This intraocular pressure elevation which lasts about 30 minutes, can result in irreversible visual loss especially in patients with critical remaining nerve fibers in the optic nerve head, as occurs in glaucomatous patients. Is there any way to prevent or even shorten this time of intraocular pressure elevation? We tried in our study to find a suitable response for a question above, so we used several anti-glaucoma agents (Timolol, Brimonidine, Acetazolamide, Mannitol versus placebo) as a prophylaxis to prevent acute intraocular pressure elevation right after intravitreal bevacizumab injection.

ELIGIBILITY:
Inclusion Criteria:

* all patients who candidate for receiving intravitreal bevacizumab

Exclusion Criteria:

* patients who had advanced glaucoma
* patients who received antiglaucoma agents in the past
* patients who had corneal scar which affect IOP measurement

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
change in IOP | 0, 5, 10, 15, 30 minutes after injection
  the change in intraocular pressure after intravitreal injection of bevacizumab

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Shoeibi, M.D., Principal Investigator — Retina Research Center, Mashhad University of Medical Sciences, Mashhad, Iran
Locations (1):
- Retina Research Center, Khatam eye Hospital, Mashhad, Khorasan Razavi, Iran

REFERENCES:
- [Derived] Shoeibi N, Ghosi Z, Jafari H, Omidtabrizi A. Effect of antiglaucoma agents on short-term intraocular pressure fluctuations after intravitreal bevacizumab injections. Int Ophthalmol. 2021 Mar;41(3):1081-1090. doi: 10.1007/s10792-020-01667-z. Epub 2021 Jan 2. PMID 33389369